CLINICAL TRIAL: NCT01450709
Title: Observational Clinical Trials of Kibow Biotics® (a Patented and Proprietary Probiotic Formulation) in Dialysis Patients, in Conjunction With Standardized Care of Treatment
Brief Title: Observational Study of Kibow Biotics in Chronic Kidney Failure Patients on Dialysis
Status: Completed | Type: Observational
Sponsor: Kibow Pharma (Industry)
Collaborators: State University of New York - Downstate Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: KIB004
Record Dates: First submitted 2011-09-26; First posted 2011-10-12 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Chronic Kidney Disease
Keywords: Probiotics; Kibow Biotics; Dialysis; Gut based uremic toxin removal
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood serum, plasma and lymphocytes.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Dialysis patients
  Interventions: Dietary Supplement: Kibow Biotics

INTERVENTIONS:
Dietary Supplement: Kibow Biotics — 6 month, double-blind, cross-over, wash-out, placebo controlled study in an outpatient setting. Each patient takes two capsules, three times a day (180 CFU/day).

SUMMARY:
A specifically formulated probiotic product comprised of defined and tested microbial strains may afford renoprotection in what has been generally called "Enteric DialysisTM". However, it is also referred to as enteric toxin reduction technology. Our hypothesis is to assess the potential benefits in devising a bowel-based probiotic formulation (Kibow® Biotics/RenadylTM) as a dietary supplement product for patients undergoing dialysis along with standardized care of treatment.

DETAILED DESCRIPTION:
Probiotics are increasingly utilized clinically. As their safety and health benefits are established, it is reasonable to anticipate that probiotic bacteria will be incorporated into a growing number of clinical regimens, as a dietary supplement.

Extensive in vitro R&D investigations in Kibow's laboratories

Bacterial strains studied were a mixture of patented and proprietary strains of Streptococcus thermophilus (KB27), Lactobacillus acidophilus (KB31) and Bifidobacterium longum (KB35).

Oral administration of these bacterial formulations, tested in the 5/6th nephrectomized rat model (at Thomas Jefferson University, Phila., PA) and minipig model (at Indiana University, Indianapolis, IN), decreased both blood urea nitrogen (BUN) and serum creatinine (Scr) levels.

Two independent veterinarians investigated the effect of Kibow Biotics® in cats and dogs (of both genders and varying body weights) with moderate to severe kidney failure. Based on positive results, this formulation, marketed and distributed as AzodylTM, is currently licensed for veterinary applications to Vetoquinol USA.

Pilot scale studies, double blind, placebo controlled, cross-over studies for six months conducted in 45 patients in USA, Canada, Argentina, and Nigeria demonstrates reduction of BUN (P>95%) and improved quality of life (P>95%). Decrease in creatinine and uric acid levels were also observed. However, these studies were based on correlating the age of geriatric cats and dogs with moderate to significant kidney failure to human geriatric conditions.

ELIGIBILITY:
Inclusion Criteria:

* Currently on hemodialysis
* 18 to 75 years of age
* Willing to give informed consent
* Baseline serum creatinine >2.5 mg/dL

Exclusion Criteria:

* Pregnant or nursing women
* Refusal to sign the informed consent form
* Documented to have HIV/AIDS/Liver disease
* Active dependency on drugs or alcohol
* Currently on anticoagulant therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Out patient hospital setting
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
15-20% Changes in BUN. | 6 months
15-20% Changes in Creatinine | 6 months
15-20% Changes in CRP | 6 months
15-20% Changes in Uric Acid Levels | 6 months

SECONDARY OUTCOMES:
Quality of life outcome based on SF 36 questionnaire. | 6 months
To observe inflammatory and oxidative stress biomarkers. | 6 months
  Observe inflammatory markers IL-1beta, NF-kappaB, Protein Bound Pentosidine, Beta2 Microglobulin, Indoxyl sulfate, Phenols, p-cresols, and guanadine metabolites from blood serum.
Observation and analysis of patient fecal matter. | 6 months
  Observation and analysis of patient fecal matter to determine bacterial flora levels that are present in the stool.

CONTACTS AND LOCATIONS:
Overall Officials: Subodh J Saggi, M.D., MPH, Principal Investigator — Downstate Medical Center; Mary Mallapallil, M.D., Principal Investigator — Kings County Medical Center; Eli Friedman, M.D., MACP, FRCP, Principal Investigator — Downstate Medical Center; Gary Briefel, M.D., Principal Investigator — Kings County Medical Center
Locations (1):
- Parkside Dialysis Clinic at Downstate Medical Center, Brooklyn, New York, United States

REFERENCES:
- [Result] Ranganathan N, Friedman EA, Tam P, Rao V, Ranganathan P, Dheer R. Probiotic dietary supplementation in patients with stage 3 and 4 chronic kidney disease: a 6-month pilot scale trial in Canada. Curr Med Res Opin. 2009 Aug;25(8):1919-30. doi: 10.1185/03007990903069249. PMID 19558344
- [Result] Ranganathan N, Ranganathan P, Friedman EA, Joseph A, Delano B, Goldfarb DS, Tam P, Rao AV, Anteyi E, Musso CG. Pilot study of probiotic dietary supplementation for promoting healthy kidney function in patients with chronic kidney disease. Adv Ther. 2010 Sep;27(9):634-47. doi: 10.1007/s12325-010-0059-9. Epub 2010 Aug 16. PMID 20721651
- [Derived] Cooper TE, Khalid R, Chan S, Craig JC, Hawley CM, Howell M, Johnson DW, Jaure A, Teixeira-Pinto A, Wong G. Synbiotics, prebiotics and probiotics for people with chronic kidney disease. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD013631. doi: 10.1002/14651858.CD013631.pub2. PMID 37870148